CLINICAL TRIAL: NCT04672655
Title: Overcoming Barriers and Obstacles to Adopting Diabetes Devices (ONBOARD) Trial
Acronym: ONBOARD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Molly Tanenbaum (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor-Investigator, Molly Tanenbaum, Clinical Assistant Professor, Stanford University
Organization: Stanford University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 56922; 1K23DK119470-01 (NIH)
Record Dates: First submitted 2020-12-11; First posted 2020-12-17 (Actual); Results first posted 2025-09-05 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-08

CONDITIONS: Type 1 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Intervention Model Description: Participants will then be randomized to receive ONBOARD or CGM-only. Those randomized to the ONBOARD condition will schedule 4 60-minute sessions with study interventionist (every 3 weeks).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- ONBOARD Intervention Group (Experimental): Those randomized to the ONBOARD group will receive 12 weeks of CGM supplies and provide hemoglobin A1c values, data downloads, and survey responses during various time points in the study. They will also receive the intervention which consists of four 60-minute sessions with study interventionist, held 2 weeks apart.
  Interventions: Behavioral: ONBOARD
- CGM Only Group (No Intervention): Those randomized to the CGM Only group will not receive the ONBOARD intervention during their 12-month participation in the study. They will only receive 12 weeks of CGM supplies and provide hemoglobin A1c values, data downloads, and survey responses during various time points in the study.

INTERVENTIONS:
Behavioral: ONBOARD — Session 1: Overview; Wearing diabetes devices; Session 2: Managing CGM data; Session 3: CGM & social situations; Session 4: Building trust with your CGM
  Arms: ONBOARD Intervention Group

SUMMARY:
This study is a comprehensive, multicomponent behavioral intervention package (ONBOARD; OvercomiNg Barriers & Obstacles to Adopting Diabetes Devices). ONBOARD will provide adults with T1D the skills to maximize benefit and minimize daily interference from barriers associated with Continuous Glucose Monitoring (CGM) and increase readiness for closed loop.

DETAILED DESCRIPTION:
The investigators will enroll 178 adults with T1D between 18-50 years of age. Participants must not have been using CGM regularly for past 6 months. Once consented and enrolled, baseline demographic and psychosocial data will be obtained. Participants will receive 12 weeks of CGM supplies at no cost to them and provided with initial standard CGM introduction and education. Participants will then be randomized to receive ONBOARD or CGM-only. Those randomized to the ONBOARD condition will schedule 4 60-minute sessions with study interventionist (every 2 weeks). Hemoglobin A1c values, CGM usage data, and psychosocial data will be collected at baseline, 3-months (post-intervention), and 6- and 12-months post-baseline.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is age 18-50 years at time of enrollment
2. Subject must not have been using CGM regularly for past 6 months
3. Subject has a clinical diagnosis of type 1 diabetes
4. Subject comprehends spoken and written English

Exclusion Criteria:

1. Subject has a medical disorder that in the judgment of the investigator will interfere with completion of any aspect of the protocol.
2. Subject has a neurologic disorder that in the judgment of the investigator will affect completion of the protocol.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 150 (Actual)
Dates: Start 2021-02-17 (Actual); Primary Completion 2024-09-16 (Actual); Study Completion 2024-09-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Molly Tanenbaum, PhD, Principal Investigator — Stanford University
Locations (1):
- Stanford University, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 150 patients signed informed consent; of these, 138 completed the baseline survey, and 135 were randomized.
Groups:
- ONBOARD Intervention Group: Those randomized to the ONBOARD group receive 12 weeks of continuous glucose monitor (CGM) supplies and provide hemoglobin A1c values, data downloads, and survey responses during various time points in the study. They also receive the intervention which consists of four 60-minute sessions with study interventionist, held 2 weeks apart.
- CGM Only Group: Those randomized to the CGM Only group do not receive the ONBOARD intervention during their 12-month participation in the study. They only receive 12 weeks of CGM supplies and provide hemoglobin A1c values, data downloads, and survey responses during various time points in the study.
Period: Overall Study
Arm/Group | ONBOARD Intervention Group | CGM Only Group
Started | 68 | 67
Met Eligibility Criteria | 67 | 67
Completed 3 Months | 61 | 60
Completed 6 Months | 57 | 54
Completed | 54 | 50
Not Completed | 14 | 17
Not completed — Lost to Follow-up | 12 | 17
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Withdrawal by Study | 1 | 0

BASELINE CHARACTERISTICS:
Population: Participants who met eligibility criteria
Groups:
- ONBOARD Intervention Group: Those randomized to the ONBOARD group receive 12 weeks of CGM supplies and provide hemoglobin A1c values, data downloads, and survey responses during various time points in the study. They also receive the intervention which consists of four 60-minute sessions with study interventionist, held 2 weeks apart.
- Total: Total of all reporting groups
Arm/Group | ONBOARD Intervention Group | CGM Only Group | Total
Number analyzed (Participants) | 67 | 67 | 134
Age, Continuous [Mean (Standard Deviation); unit: years] | 34.50 (8.87) | 34.86 (7.92) | 34.68 (8.38)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 54 | 49 | 103
  Male | 13 | 17 | 30
  Non-binary | 0 | 1 | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 5 | 4 | 9
  Black or African American | 2 | 3 | 5
  Hispanic/Latinx | 5 | 1 | 6
  Native Hawaiian/Pacific Islander | 1 | 0 | 1
  White | 49 | 52 | 101
  Other | 0 | 2 | 2
  More than one | 5 | 5 | 10
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 67 | 67 | 134
Hemoglobin A1c (HbA1c) [Mean (Standard Deviation); unit: Percentage of Glycated Hemoglobin] | 8.20 (1.78) | 7.85 (1.96) | 8.03 (1.87)
Diabetes Distress Scale for Adults With Type 1 Diabetes (T1-DDS) [Mean (Standard Deviation); unit: Score on a scale] — The T1-DDS is a 28-item self-report scale that assesses multiple dimensions of diabetes distress. Each item is scored from 1 to 6, then items scores are summed and average to calculate a total score (1 to 6). Higher item and total scores indicate more distress (worse outcome).
  Score on a scale | 2.5 (0.87) | 2.48 (0.82) | 2.49 (0.84)
Percent Time in Glucose Target Range [Mean (Standard Deviation); unit: Percentage of time] — This characteristic was assessed for 2 weeks prior to the baseline visit.
  Percentage of time | 0.58 (0.19) | 0.61 (0.2) | 0.59 (0.19)
Percent CGM Wear Time [Mean (Standard Deviation); unit: Percentage of time] — This characteristic was assessed for 2 weeks prior to the baseline visit.
  Percentage of time | 12.28 (2.09) | 12.18 (2.01) | 12.23 (2.04)
Glucose Monitoring System Satisfaction Survey - Version: Type 1 Diabetes (GMSS-T1D) [Median (Standard Deviation); unit: Score on a scale] — The GMSS-T1D is a 15-item self-report scale that assesses attitudes towards one's current glucose monitoring system. Each item is scored from 1 to 5, then items scores are summed and average to calculate a total score (1 to 5). Higher item and total scores indicate greater satisfaction (better outcome).
  Score on a scale | 3.31 (0.63) | 3.19 (0.62) | 3.25 (0.63)

OUTCOME MEASURES:

1. Primary Outcome: Change in Hemoglobin A1c (HbA1c) Over Time
Description: Glycated hemoglobin
Time Frame: baseline, month 3, month 6, month 12
Population: Participants with data at each respective time point
Measure: Least Squares Mean (95% Confidence Interval); unit: percentage of glycated hemoglobin
Arm/Group | ONBOARD Intervention Group | CGM Only Group
Number analyzed (Participants) | 53 | 57
percentage of glycated hemoglobin
  Change at Month 3 | -0.34 [-0.61 to -0.06] | -0.53 [-0.80 to -0.26]
  Change at Month 6: number analyzed (Participants) | 44 | 51
  Change at Month 6 | -0.34 [-0.61 to -0.06] | -0.51 [-0.79 to -0.23]
  Change at Month 12: number analyzed (Participants) | 53 | 49
  Change at Month 12 | -0.21 [-0.49 to -0.07] | -0.48 [-0.76 to -0.19]
Statistical Analysis 1: Comparison: ONBOARD Intervention Group vs CGM Only Group; A linear mixed effects model (LMM) was used to examine outcomes measured at 3, 6, and 12 months. An unstructured covariance matrix was specified to model within-subject correlations across repeated measurements. To address missing data, the LMM utilized a likelihood-based approach under the missing-at-random (MAR) assumption, which incorporates all available data, thereby minimizing bias from incomplete follow-up measurements; Test type: Other; p = 0.8875, linear mixed effects models — The a priori threshold for statistical significance was < 0.05

2. Secondary Outcome: Change in Time in Glucose Target Range
Description: 14 days of CGM data were used to calculate the change in the percentage glucose readings from CGM system between 70-180 mg/dL per unit of time at each time point. All time points taken together are needed to evaluate this outcome measure.
Time Frame: baseline, month 3, month 6, month 12
Population: Participants with data at each respective time point
Measure: Least Squares Mean (95% Confidence Interval); unit: percentage of time in range
Arm/Group | ONBOARD Intervention Group | CGM Only Group
Number analyzed (Participants) | 51 | 57
percentage of time in range
  Change at month 3 | -0.03 [-0.07 to 0.01] | -0.02 [-0.05 to -0.02]
  Change at month 6: number analyzed (Participants) | 40 | 33
  Change at month 6 | -0.04 [-0.08 to 0.00] | -0.01 [-0.05 to 0.04]
  Change at month 12: number analyzed (Participants) | 35 | 30
  Change at month 12 | -0.03 [-0.07 to -0.01] | 0.00 [-0.04 to 0.05]
Statistical Analysis 1: Comparison: ONBOARD Intervention Group vs CGM Only Group; [analysis description as in outcome 1, analysis 1]; Test type: Other; p = 0.4811, linear mixed effects models — The a priori threshold for statistical significance was < 0.05

3. Secondary Outcome: Change in Percent CGM Wear Time
Description: 14 days of CGM data were used to calculate the change in percentage of time wearing CGM at each time point. All time points taken together are needed to evaluate this outcome measure.
Time Frame: baseline, month 3, month 6, month 12
Population: Participants with data at each respective time point
Measure: Least Squares Mean (95% Confidence Interval); unit: percentage of days wearing CGM
Arm/Group | ONBOARD Intervention Group | CGM Only Group
Number analyzed (Participants) | 51 | 57
percentage of days wearing CGM
  Change at Month 3 | -0.08 [-0.14 to -0.03] | -0.11 [-0.16 to -0.05]
  Change at Month 6: number analyzed (Participants) | 40 | 33
  Change at Month 6 | -0.04 [-0.11 to 0.02] | -0.07 [-0.14 to 0.00]
  Change at Month 12: number analyzed (Participants) | 34 | 30
  Change at Month 12 | -0.01 [-0.08 to 0.06] | -0.07 [-0.14 to 0.00]
Statistical Analysis 1: Comparison: ONBOARD Intervention Group vs CGM Only Group; [analysis description as in outcome 1, analysis 1]; Test type: Other; p = 0.754, linear mixed effects models — The a priori threshold for statistical significance was < 0.05

4. Secondary Outcome: Change in Diabetes Distress Scale for Adults With Type 1 Diabetes (T1-DDS)
Description: The T1-DDS is a 28-item self-report scale that assesses multiple dimensions of diabetes distress. Each item is scored from 1 to 6, then items scores are summed and average to calculate a total score (1 to 6): higher item and total scores indicate more distress (worse outcome). All time points taken together are needed to evaluate this outcome measure
Time Frame: baseline, month 3, month 6, month 12
Population: Participants with data at each respective time point
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | ONBOARD Intervention Group | CGM Only Group
Number analyzed (Participants) | 67 | 67
score on a scale
  Change at Month 3: number analyzed (Participants) | 58 | 58
  Change at Month 3 | -0.24 [-0.39 to -0.10] | -0.48 [-0.63 to -0.34]
  Change at Month 6: number analyzed (Participants) | 52 | 15
  Change at Month 6 | -0.32 [-0.47 to -0.17] | -0.39 [-0.54 to -0.24]
  Change at Month 12: number analyzed (Participants) | 54 | 16
  Change at Month 12 | -0.38 [-0.53 to -0.23] | -0.38 [-0.53 to -0.23]
Statistical Analysis 1: Comparison: ONBOARD Intervention Group vs CGM Only Group; [analysis description as in outcome 1, analysis 1]; Test type: Other; p = 0.0406, linear mixed effects models — The a priori threshold for statistical significance was < 0.05

5. Secondary Outcome: Change in Glucose Monitoring System Satisfaction Survey - Version: Type 1 Diabetes (GMSS-T1D)
Description: The GMSS-T1D is a 15-item self-report scale that assesses attitudes towards one's current glucose monitoring system. Overall score range is 1 to 5: higher total scores indicate greater satisfaction (better outcome). All time points taken together are needed to evaluate this outcome measure
Time Frame: baseline, month 3, month 6, month 12
Population: Participants with data at each respective time point
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | ONBOARD Intervention Group | CGM Only Group
Number analyzed (Participants) | 58 | 58
score on a scale
  Change at Month 3 | 0.61 [0.46 to 0.76] | 0.53 [0.38 to 0.69]
  Change at Month 6: number analyzed (Participants) | 52 | 52
  Change at Month 6 | 0.5 [0.34 to 0.66] | 0.47 [0.32 to 0.63]
  Change at Month 12: number analyzed (Participants) | 55 | 51
  Change at Month 12 | 0.47 [0.32 to 0.63] | 0.41 [0.25 to 0.57]
Statistical Analysis 1: Comparison: ONBOARD Intervention Group vs CGM Only Group; [analysis description as in outcome 1, analysis 1]; Test type: Other; p = 0.9032, linear mixed effects models — The a priori threshold for statistical significance was < 0.05

ADVERSE EVENTS:
Time Frame: Up to 12 months
Arm/Group | ONBOARD Intervention Group | CGM Only Group
All-Cause Mortality (participants affected / at risk) | 0/68 | 0/67
Serious Adverse Events (participants affected / at risk) | 4/68 | 1/67
Other Adverse Events (participants affected / at risk) | 0/68 | 0/67
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | ONBOARD Intervention Group (N=68) | CGM Only Group (N=67)
Vomiting (Gastrointestinal disorders) | 1 | 0 — Unrelated to study participation.
Appendicitis (Surgical and medical procedures) | 1 | 0 — Unrelated to study participation.
Diabetic Ketoacidosis (Endocrine disorders) | 1 | 1 — Unrelated to study participation.
Hypoglycemic Episode (Endocrine disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-11-11): https://cdn.clinicaltrials.gov/large-docs/55/NCT04672655/Prot_SAP_002.pdf
  • Informed Consent Form (2024-07-16): https://cdn.clinicaltrials.gov/large-docs/55/NCT04672655/ICF_001.pdf